CLINICAL TRIAL: NCT06246669
Title: The Influence of Prescribed Exercise on Pain Related Fear Following Concussion in Collegiate Athletes: A Randomized Controlled Trial
Brief Title: The Influence of Prescribed Exercise on Pain Related Fear Following Concussion in Collegiate Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jacob Resch, Associate Professor, Department of Kinesiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR230522
Record Dates: First submitted 2024-01-20; First posted 2024-02-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Concussion, Brain
Keywords: kinesiophobia; exercise; anxiety
MeSH Terms: conditions — Brain Concussion; Kinesiophobia; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity (Experimental): Treadmill walking at a rating of perceived exertion (RPE) of 13.
  Interventions: Behavioral: Treadmill Walking
- Light Intensity (Experimental): Treadmill walking at a rating of perceived exertion (RPE) of 9.
  Interventions: Behavioral: Treadmill Walking

INTERVENTIONS:
Behavioral: Treadmill Walking — A treadmill will be used for participant to walk on. The frequency of exercise will be 5 times per week until they report symptom-free. The intensity will be determined via random group allocation (RPE of 13 or 9). The type of exercise is treadmill walking. The time of the intervention will depend on the the time it takes an individual to reach a specific caloric expenditure as a function of their weight and treadmill incline. This is based on the most recent American Congress of Sports Medicine's guidelines for estimating gross energy expenditure during common physical activities.

SUMMARY:
The goal of this clinical trial is to compare the effects of acute aerobic exercise at two different intensities on psychological measures, symptomology, and time to symptom free in collegiate student athletes with concussion. The main questions it aims to answer are:

* Does prescribed, acute aerobic exercise influence measures of pain related fear, anxiety, depression, symptoms, and recovery time?
* Does the intensity of the exercise prescription also influence the aforementioned outcomes?

Participants will be randomly assigned into either a light intensity or moderate intensity aerobic exercise (treadmill walking) group. They will initiate the exercise protocol 48 hours following their concussion diagnosis, and complete exercise sessions 5 times per week until they report symptom-free. Researchers will compare the light intensity group to the moderate intensity group to see if intensity of exercise influences psychological measures of pain related fear, anxiety, depression, symptomology, and time to symptom-free.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate athlete (varsity)
* Symptomatic at time of exercise prescription

Exclusion Criteria:

* If advanced neuroimaging was performed, any subject with a structural abnormality will be excluded
* History of traumatic brain injury requiring hospitalization
* Not cleared to play their sport by a physician due to some other injury such as an ankle sprain or muscle strain
* If individual is diagnosed with any condition that is a contraindication to aerobic exercise. Please note that all participants will have already been cleared to participate in their respective collegiate sport after extensive pre-participation physical examinations upon entering the university.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The Tampa Scale of Kinesiophobia-17 (TSK-17) | 48 hours after concussion diagnosis and then every other day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  A measure of fear beliefs associated with exercise, movement, and re-injury. Minimum score of 17, Maximum 68. Higher scores indicate worse kinesiophobia.
Athlete Fear Avoidance Questionnaire (AFAQ) | 48 hours after concussion diagnosis and then every other day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  A measure of fear avoidance specifically designed for injured athletes. Minimum score of 10, Maximum score of 50. Higher scores indicate higher levels of fear-avoidance.
Revised Head Injury Scale (HIS-r) | 48 hours after concussion diagnosis and then every single day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  A measure of 22 concussion related symptoms and their associated duration and severity over the previous 24 hours. Minimum duration of 1 and a maximum duration of 132. Minimum severity of 0 and maximum severity of 132. Higher levels of symptom count, duration, and severity indicate worse symptomology.
Days until symptom-free | Depends on individual injury characteristics but has a median of 6 days, range of 0-203 days at the research site.
  The time it takes, in days, for a participant to report symptom free.

SECONDARY OUTCOMES:
Generalized Anxiety Index-7 (GAD-7) | 48 hours after concussion diagnosis and then every other day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  Measure of anxiety levels over previous two weeks. Minimum score of 0 and maximum score of 21. Higher scores indicating higher levels of anxiety.
Patient Health Questionnaire-9 (PHQ-9) | 48 hours after concussion diagnosis and then every other day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  Measure of depression levels over previous two weeks. Minimum score of 0 and maximum score of 27. Higher scores indicate higher levels of depression.
Days until return to sport | Depends on individual injury characteristics but will be, on median, 5 days after reporting symptom free which takes 6 days on median at the research site.
  The time it takes, in days, for a participant to make a full return to their sport.
Step count | Step count recording will begin 48 hours after concussion diagnosis and then every single day until participant reports symptom free which takes, on median, 6 days with a range of 0-203 days at the research site.
  Number of steps taken during daily life outside of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia Department of Kinesiology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be available upon reasonable request from qualified individuals.
Supporting Information: Study Protocol
Time Frame: Upon study completion. Will be available indefinitely.
Access Criteria: Data will be available upon reasonable request from qualified individuals.

REFERENCES:
- [Background] Leddy JJ, Burma JS, Toomey CM, Hayden A, Davis GA, Babl FE, Gagnon I, Giza CC, Kurowski BG, Silverberg ND, Willer B, Ronksley PE, Schneider KJ. Rest and exercise early after sport-related concussion: a systematic review and meta-analysis. Br J Sports Med. 2023 Jun;57(12):762-770. doi: 10.1136/bjsports-2022-106676. PMID 37316185
- [Background] Lal A, Kolakowsky-Hayner SA, Ghajar J, Balamane M. The Effect of Physical Exercise After a Concussion: A Systematic Review and Meta-analysis. Am J Sports Med. 2018 Mar;46(3):743-752. doi: 10.1177/0363546517706137. Epub 2017 Jun 1. PMID 28570092
- [Background] Lawrence DW, Richards D, Comper P, Hutchison MG. Earlier time to aerobic exercise is associated with faster recovery following acute sport concussion. PLoS One. 2018 Apr 18;13(4):e0196062. doi: 10.1371/journal.pone.0196062. eCollection 2018. PMID 29668716
- [Background] Thompson XD, Newman TM, Donahue CC, Erdman NK, Statuta SM, Resch JE. Kinesiophobia Is Related to Acute Musculoskeletal Injury Incidence Following Concussion. J Sport Rehabil. 2022 Sep 1;32(2):145-150. doi: 10.1123/jsr.2022-0134. Print 2023 Feb 1. PMID 36049743
- [Background] Reinking S, Seehusen CN, Walker GA, Wilson JC, Howell DR. Transitory kinesiophobia after sport-related concussion and its correlation with reaction time. J Sci Med Sport. 2022 Jan;25(1):20-24. doi: 10.1016/j.jsams.2021.07.010. Epub 2021 Jul 29. PMID 34404602
- [Background] Jadhakhan F, Sobeih R, Falla D. Effects of exercise/physical activity on fear of movement in people with spine-related pain: protocol for a systematic review and meta-analysis. BMJ Open. 2022 May 19;12(5):e060264. doi: 10.1136/bmjopen-2021-060264. PMID 35589367
- [Background] Patricios JS, Schneider KJ, Dvorak J, Ahmed OH, Blauwet C, Cantu RC, Davis GA, Echemendia RJ, Makdissi M, McNamee M, Broglio S, Emery CA, Feddermann-Demont N, Fuller GW, Giza CC, Guskiewicz KM, Hainline B, Iverson GL, Kutcher JS, Leddy JJ, Maddocks D, Manley G, McCrea M, Purcell LK, Putukian M, Sato H, Tuominen MP, Turner M, Yeates KO, Herring SA, Meeuwisse W. Consensus statement on concussion in sport: the 6th International Conference on Concussion in Sport-Amsterdam, October 2022. Br J Sports Med. 2023 Jun;57(11):695-711. doi: 10.1136/bjsports-2023-106898. PMID 37316210